CLINICAL TRIAL: NCT01216046
Title: A Phase 1, Randomized, Double-Blind, Placebo Controlled, Multiple-Dose, Dose-Escalation, Drug-Drug Interaction Study of VX-809 and VX-770 in Healthy Subjects
Brief Title: Drug-Drug Interaction Study of VX-770 and VX-809 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX10-809-006
Record Dates: First submitted 2010-09-29; First posted 2010-10-07 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm (Experimental): Subjects randomized to study drug will take VX-809 for 14 days followed by a 14 day washout. Next subjects will take VX-770 for 14 days followed by a 14 day washout. Lastly, subjects will take both VX-809 and VX-770 for 14 days.
  Interventions: Drug: VX-809; Drug: VX-770
- Placebo Arm (Placebo Comparator): Subjects randomized to placebo will take VX-809 placebo for 14 days followed by a 14 day washout. Next subjects will take VX-770 placebo for 14 days followed by a 14 day washout. Lastly, subjects will take both VX-809 and VX-770 placebo for 14 days.
  Interventions: Drug: VX-809 placebo; Drug: VX-770 placebo

INTERVENTIONS:
Drug: VX-809 — capsule, taken once daily
  Arms: Treatment Arm
Drug: VX-770 — tablet, taken once every 12 hours
  Arms: Treatment Arm
Drug: VX-809 placebo — capsule, taken once daily
  Arms: Placebo Arm
Drug: VX-770 placebo — tablet, taken once every 12 hours
  Arms: Placebo Arm

SUMMARY:
The purpose of this study is to assess the pharmacokinetics and safety of VX-809 and VX-770 alone and in combination in healthy subjects.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, multiple-dose study of orally administered VX-809 and VX-770 in healthy subjects. This study will evaluate safety and tolerability of VX-809 and VX-770 alone and in combination.

Subjects will be randomized to receive study drug or placebo during three 14-day treatment periods separated by 14-day washout periods. In Treatment Period 1, subjects randomized to study drug will receive VX-809 every 24 hours. In Treatment Period 2, subjects randomized to study drug will receive VX-770 every 12 hours. In Treatment Period 3, subjects will receive VX-809 every 24 hours and VX-770 every 12 hours. Subjects randomized to placebo will receive placebo during all treatment periods.

Enrollment is planned at 1 clinical site (Lenexa, Kansas). Up to 72 subjects will be enrolled. The study will be separated into 3 dose escalation cohorts. Cohort 1 and Cohort 2 will enroll 24 subjects. Cohort 3 is optional and may be conducted after a review of safety and pharmacokinetic data by Vertex.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject between 18 and 55 years of age, inclusive
* Body mass index (BMI) between 18.5 and 30.0 kg/m2, inclusive
* Subjects of child bearing potential and who are sexually active must meet the contraception requirements
* Female subject must have a negative serum pregnancy test at screening and Day -1

Exclusion Criteria:

* History of any illness that, in the opinion of the investigator might confound the results of the study or pose an additional risk in administering study drug to the subject
* Participated in a clinical study involving administration of either an investigational or a marketed drug within 30 days or 5 terminal half-lives (whichever is longer) before the Screening visit
* Subject who has received VX-770 or VX-809 in a previous clinical study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
PK parameters (including concentration, exposure and half-life) of VX-809 and its metabolite in plasma in the presence and absence of VX 770 | 70 days
  Blood samples drawn during the study will be analyzed to measure the PK parameters, such as concentration, exposure and half-life of VX-809 and its metabolite.
PK parameters (including concentration, exposure and half-life) of VX-770 and its metabolites in plasma in the presence and absence of VX 809 | 70 days
  Blood samples drawn during the study will be analyzed to measure the PK parameters, such as concentration, exposure and half-life of VX-770 and its metabolites.

SECONDARY OUTCOMES:
Safety and tolerability as measured by adverse events (AEs) and clinically significant changes in laboratory values (clinical chemistry, hematology, coagulation, and urinalysis), electrocardiograms, and vital signs | 70 days

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Vernillet, PharmD, PhD, FCP, Study Director — Vertex Pharmaceuticals Incorporated
Locations (1):
- PRA, Lenexa, Kansas, United States